CLINICAL TRIAL: NCT00826475
Title: Randomized Trial to Evaluate the Effectiveness of a Mindfulness Based Intervention (MBSR) for Patients Suffering From Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. Stefan Schmidt, Institute of Environmental Health Sciences, University Medical Center Freiburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 423/08
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2009-01

CONDITIONS: Migraine
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental): Mindfulness Based Stress Reduction: 8 weeks behavioral structured group programme teaching mindfulness skills
  Interventions: Behavioral: Mindfulness Based Stress Reduction MBSR
- Psychoeducation (Active Comparator): Psychoeducation on Migraine, Progressive Muscle Relaxation PMR, three group meetings within 8 weeks, daily home work
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction MBSR — Mindfulness Based Stress Reduction: 8 weeks behavioral structured group programme teaching mindfulness skills
  Arms: Mindfulness
Behavioral: Psychoeducation — Psychoeducation on Migraine, Progressive Muscle Relaxation PMR, three group meetings within 8 weeks, daily home work
  Arms: Psychoeducation

SUMMARY:
Patients suffering from migraine will be randomly allocated to one of two different behavioral interventions:

* mindfulness based stress reduction (MBSR) an eight week intervention program based different meditation & yoga techniques and teaching information regarding the relationship between stress and health.
* into an active control group teaching three times within eight weeks relaxation techniques (progressive muscle relaxation PMR) and giving psychoeducation on migraine. The investigators will measure the frequency and intensity of migraine attacks before during and after the intervention as well as secondary variables on quality of life and psychological functioning. The hypothesis is that patients allocated to the MBSR intervention will reduce the frequency of their migraine attacks compared to the active control group and compared to their own baseline.

DETAILED DESCRIPTION:
Sixty patients suffering from migraine will be randomly allocated to one of two different behavioral interventions: (i) mindfulness based stress reduction (MBSR) an eight week intervention program based different meditation & yoga techniques and teaching information regarding the relationship between stress and health. or (ii) into an active control group teaching three times within eight weeks relaxation techniques (progressive muscle relaxation PMR) and giving psychoeducation on migraine. The investigator will measure the frequency and intensity of migraine attacks before during and after the intervention by headache diaries as well as secondary variables on pain sensation, psychological well being, generic quality of life, pain regulation, pain acceptance, mindfulness, compliance and satisfaction with the intervention. The hypothesis is that patients allocated to the MBSR intervention will reduce the frequency of their migraine attacks compared to the active control group and compared to their own baseline.

ELIGIBILITY:
Inclusion Criteria:

* migraine for at least 6 months
* commandment of German language
* 3-8 migraine attacks per month
* willingness to participate in a behavioral intervention and to conduct the daily homework
* if patients take a drug as prophylaxis for migraine no change of drug for at least three months and no change of dose for at least one month prior to enrollment

Exclusion Criteria:

* psychiatric disorders at the time of enrollment
* addiction
* participation in other trials
* prior experience with mbsr
* migraine related to the ovary cycle
* abuse of acute medication for migraine
* other psychological disorders which impair the communication and interaction with the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
number of days suffering from migraine-type headache per month to be determined by a headache diary | one month

SECONDARY OUTCOMES:
pain sensation scale (Schmerzempfindungsskala) | at post intervention
Brief Symptom Inventory (BSI) | post intervention
Freiburg Mindfulness Inventory (FMI) | post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany